CLINICAL TRIAL: NCT04840914
Title: A Single-Dose Study Evaluating Different Dose Levels and Subcutaneous Infusion Durations on Safety, Pharmacokinetics, and Pharmacodynamics of LY3461767 in Participants With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: A Study of LY3461767 in Participants With Chronic Heart Failure With Reduced Ejection Fraction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17518; J2L-MC-EZBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-09; First posted 2021-04-12 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3461767 (Experimental): LY3461767 administered subcutaneously (SC).
  Interventions: Drug: LY3461767
- Placebo (Placebo Comparator): Placebo administered subcutaneously (SC).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3461767 — Administered SC.
  Arms: LY3461767
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the tolerability and safety of LY3461767 with any side effects that might be associated with it. Study drug will be provided in a continuous subcutaneous infusion lasting 24 hours to 96 hours, depending on the cohort. Blood tests will be performed to check concentrations of LY3461767 in the bloodstream and how long it takes the body to get rid of it in participants with chronic heart failure with reduced ejection fraction (HFrEF). The study will last up to 3 months and may include 5 visits.

ELIGIBILITY:
Inclusion Criteria:

* Are males and in agreement to follow contraceptive requirements, or women of non-child-bearing potential
* Have a body mass index (BMI) of </= 45.0 kilograms per square meter (kg/m²)
* Have chronic stable heart failure (New York Heart Association (NYHA) classification II and III) on guideline directed heart failure therapy for at least 6 months prior to enrolment
* Have not changed optimal guideline directed therapy in the last 1 month prior to screening, If treated with oral diuretics, dose must be stable for at least 2 weeks prior to screening
* Have Left Ventricular Ejection Fraction (LVEF) < 40%
* Have a record of N-terminal pro b-type natriuretic peptide (NT-ProBNP) ≥ 200 picograms per millilitre (pg/mL) or a BNP value of >/= 60 pg/mL within the past 12 months prior to screening

Exclusion Criteria:

* Have myocardial infarction, coronary artery bypass graft surgery or other major cardiovascular surgery, stroke in the last 90 days prior to screening
* Have acute decompensated heart failure requiring IV diuretics within 12 weeks prior to screening
* Have cardiac amyloidosis, accumulation diseases (e.g., haemochromatosis, Fabry disease), muscular dystrophies, hypertrophic cardiomyopathy, pericardial constriction, or complex congenital heart disease.
* Have any moderate-to-severe stenosis of the mitral and/or aortic valve or moderate-to severe or greater mitral and/or aortic regurgitation.
* Have a history or presence of hepatic, pancreatic, or biliary tract disorders
* Have a history of malignancy or active malignancy at screening.
* Have not had age-appropriate cancer screening as recommended by the American Cancer Society and per medical judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 90
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3461767 | Predose up to 48 hours post end of infusion
  PK: AUC of LY3461767
PK: Maximum Concentration (Cmax) of LY3461767 | Predose up to 48 hours post end of infusion
  PK: Cmax of LY3461767

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (3):
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - University of North Carolina, Division of Cardiology, Chapel Hill, North Carolina
- Japan (4):
  - Tsuchiura Kyodo Hospital, Tsuchiura, Ibaraki
  - Kanagawa Prefectural Hospital Organization Kanagawa Cardiovascular and Respiratory Center, Kanazawa Ward,Yokohama, Kanagawa
  - National Cerebral and Cardiovascular Center, Suita-shi, Osaka
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3461767 in Participants With Chronic Heart Failure With Reduced Ejection Fraction — https://trials.lillytrialguide.com/en-US/trial/1W0ItmrE6ruLINUYr7X1m5